CLINICAL TRIAL: NCT07167173
Title: Predictive Model for Multidrug Resistance in Patients Admitted to the Emergency Department With Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, EMILIO FELIPE HUAIER ARRIAZU, Infectious disease physician, member of the Infectious disease department and the Infection control committee of Hospital Italiano de Buenos Aires, Hospital Italiano de Buenos Aires
Other Study IDs: 7441
Record Dates: First submitted 2025-07-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sepsis; Septic Shock
Keywords: Antimicrobial resistance; sepsis; predictive models
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with sepsis: Individuals aged 18 years or older who present to the Adult Emergency Department (CEA) at the Hospital Italiano de Buenos Aires between 01/01/2017 and 10/08/2025 with sepsis or septic shock and requiring at least 48 hours of observation or admission. The COVID-19 pandemic period will be excluded.

SUMMARY:
Introduction: Timely and accurate antibiotic administration in emergency department (ED) patients with sepsis or septic shock is vital, given mortality rates of 20% and over 40%, respectively. In high antimicrobial resistance (AMR) settings, selecting effective empirical antibiotics is challenging, requiring a balance between efficacy and minimizing multidrug-resistant organism (MDRO) emergence. A predictive model estimating AMR probability could optimize antibiotic use, improve outcomes, and reduce resistance. Although risk factors are known, no single validated model exists for predicting multidrug resistance in sepsis. Accurate prediction must integrate patient history, pathogen profiles, infection source, and antibiotic characteristics.

Objectives: To estimate AMR prevalence in adult ED patients with sepsis or septic shock and develop a validated predictive model estimating AMR probability and likely pathogens. The model will follow a three-phase approach: (1) predict culture positivity, (2) estimate pathogen likelihood, and (3) predict AMR. Additionally, we aim to describe individual-level statistics for both predictable and unpredictable cases based on model performance.

Methods: A cross-sectional study will be conducted at Hospital Italiano's adult ED over 70 months (Jan 1, 2017-Mar 20, 2020 and May 1, 2022-Aug 10, 2025), excluding the COVID-19 period. Primary outcomes include culture positivity, bacterial species, and MDRO prevalence. Frequency analyses will use positive cultures, species, and resistance classifications (MDRO, MDR, XDR, PDR), including mechanisms (e.g., MRSA, ESBL, KPC, MBL, OXA). Denominators will include all sepsis patients and, separately, culture-positive cases. Confidence intervals (95%) will be calculated using normal approximation. Multivariate logistic regression with backward stepwise selection will identify predictors and interactions. A hierarchical model will be developed based on culture results, pathogen identification, and resistance profiles.

DETAILED DESCRIPTION:
Introduction:

Timely and accurate antibiotic administration in emergency department (ED) patients with sepsis or septic shock is vital, given mortality rates of 20% and over 40%, respectively. In high antimicrobial resistance (AMR) settings, selecting effective empirical antibiotics is challenging, requiring a balance between efficacy and minimizing multidrug-resistant organism (MDRO) emergence. A predictive model estimating AMR probability could optimize antibiotic use, improve outcomes, and reduce resistance. Although risk factors are known, no single validated model exists for predicting multidrug resistance in sepsis. Accurate prediction must integrate patient history, pathogen profiles, infection source, and antibiotic characteristics.

Objectives

In adult patients who present to an emergency department in a tertiary care center with sepsis or septic shock:

1-Prevalence and Associated Factors

1a- Estimate the prevalence of AMR/resistance patterns with clinical significance.

1b- Describe the predictive factors associated with AMR in this population.

1c- Generally, and in clinically relevant subgroups: by probable focus, clinically relevant pathogens, severity.

2- Generation and Validation of Predictive Models 2a- Generate and validate clinically useful predictive models to predict the probability of AMR.

2b- Generate and validate clinically useful predictive models to predict the probability of common/relevant pathogens.

2c- Evaluate the performance of stepwise predictive models in three stages: 1. Prediction of positive culture, 2. Intermediate prediction of pathogen, and 3. Prediction of AMR.

2d- Describe and evaluate point statistics on deterministic and unpredictable individuals based on the best predictive models.

Methods:

A cross-sectional study will be conducted at Hospital Italiano's adult ED over 70 months (Jan 1, 2017-Mar 20, 2020 and May 1, 2022-Aug 10, 2025), excluding the COVID-19 period. Primary outcomes include culture positivity, bacterial species, and MDRO prevalence. Frequency analyses will use positive cultures, species, and resistance classifications (MDRO, MDR, XDR, PDR), including mechanisms (e.g., MRSA, ESBL, KPC, MBL, OXA). Explanatory variables - Potential predictors of resistance include: Patient characteristics, Invasive devices, Immunosuppression, Comorbidities, Therapeutic adequacy, Medical history, Antibiotic use, Clinical status and Diagnostic studiesDenominators will include all sepsis patients and, separately, culture-positive cases. Confidence intervals (95%) will be calculated using normal approximation. Multivariate logistic regression with backward stepwise selection will identify predictors and interactions.

A hierarchical model will be developed based on culture results, pathogen identification, and resistance profiles. The sample will be randomly divided into a generation sample (2/3 of the sample) and a validation sample (1/3 of the sample). For the generation and validation of predictive models, the positive culture, each selected relevant bacteria, MDRO, MDR, XDR, PDR will be used as outcome variables.

List of Abbreviations (Abbreviation - Meaning) ABA - Acinetobacter baumannii AMR - Antimicrobial Resistance ESBL - Extended Spectrum Beta-Lactamase-producing Enterobacterales ESKAPE - Acronym summarizing the main clinically relevant resistant germs currently, each letter represents the initial of the scientific name of the bacterium: Enterococcus faecium, Staphylococcus aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa, Enterobacter spp.

CPE - carbapenemase-producing Enterobacteriaceae GNB - Gram-Negative Bacilli GPC - Gram-Positive Cocci KPC - Carbapenem-resistant Klebsiella pneumoniae MBL - Metallo-beta-lactamase MDR - Multidrug-resistant MOR - Multidrug-resistant Organisms MRSA - Methicillin-resistant Staphylococcus aureus OXA - Oxacillinase-type Carbapenemase PAE MR - Multidrug-resistant Pseudomonas aeruginosa PDR - Pan-resistant SOFA - Sepsis-related Organ Failure Assessment SSC - Surviving Sepsis Campaign VRE - Vancomycin-resistant Enterococci XDR - Extremely resistant

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older.
* Attended at the Adult Emergency Department of Hospital Italiano de Buenos Aires during the periods:

  * January 1, 2017 - March 20, 2020, or
  * May 1, 2022 - August 10, 2025.
* Sepsis or septic shock at presentation and at least 48 hours of observation or hospital admission.
* Bacterial cultures obtained during the initial evaluation.

Exclusion Criteria

* No indication for antibiotic therapy within the first 48 hours of hospital admission.
* No bacterial cultures performed within the first 48 hours of hospital admission.
* SARS-CoV-2 infection diagnosed within the first 72 hours of hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 years or older with sepsis.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of episodes with multidrug-resistant organisms (MDRO) | Baseline (within the first 48 hours of admission)
  Percentage of episodes with a positive bacterial culture that meet criteria for multidrug resistance (MDR or greater, i.e., MDR/XDR/PDR), defined according to Magiorakos et al., 2012.
  Unit of Measure: % of culture-positive episodes

SECONDARY OUTCOMES:
Culture positivity | Baseline
  Dichotomous variable. It will be considered positive or negative.
Bacterial species (Number of Participants with each microorganism species) | Baseline
  Categorical variable; the following will be considered:
  Escherichia coli, Salmonella, Shigella, Klebsiella pneumoniae, Proteus mirabilis, other Proteus species (P. penneri or P. vulgaris), Morganella morganii, Providencia stuartii, Providencia rettgeri, Serratia marcescens, Citrobacter koseri, Citrobacter freundii, Enterobacter cloacae, Klebsiella aerogenes, Hafnia alvei, Pseudomonas aeruginosa, Acinetobacter baumannii, Stenotrophomonas maltophilia, Enterococcus faecalis, Enterococcus faecium, Staphylococcus aureus, coagulase-negative Staphylococcus, Streptococcus pneumoniae, group A beta-hemolytic Streptococcus, Streptococcus pyogenes, Haemophilus influenzae, Neisseria meningitidis, Listeria monocytogenes, others.
Enzymatic resistance mechanisms (Number of Participants with each enzymatic mechanism detected) | Baseline
  Categorical variable, the following will be considered: No enzymatic mechanism; MRSA; VRE; KPC; MBL; OXA.
Carbapenemase genotypes (Number of participants with each genotypic resistance mechanism -KPC, NDM, VIM, OXA-48, IMP- detected by multiplex PCR assay) | Baseline
  Categorical variable; the following will be considered: Types of carbapenemases if studied (for example, KPC, NDM, VIM, IMP, OXA-48 like).
Proportion of episodes with MDR organisms | Baseline
  Percentage of culture-positive episodes classified as MDR (resistant to ≥1 agent in ≥3 antimicrobial categories).
  Unit of Measure: % of culture-positive episodes
Proportion of episodes with XDR organisms | Baseline
  Percentage of culture-positive episodes classified as XDR (non-susceptible to ≥1 agent in all but ≤2 categories).
  Unit of Measure: % of culture-positive episodes
Proportion of episodes with PDR organisms | Baseline
  Percentage of culture-positive episodes classified as PDR (non-susceptible to all agents in all categories).
  Unit of Measure: % of culture-positive episodes

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Felipe H Huaier Arriazu, MD, Principal Investigator — Hospital Italiano de Buenos Aires

IPD SHARING:
Plan to Share IPD: No
Not possible due to confidentiality and legal restrictions.

REFERENCES:
- [Background] Jung K, Kashyap S, Avati A, Harman S, Shaw H, Li R, Smith M, Shum K, Javitz J, Vetteth Y, Seto T, Bagley SC, Shah NH. A framework for making predictive models useful in practice. J Am Med Inform Assoc. 2021 Jun 12;28(6):1149-1158. doi: 10.1093/jamia/ocaa318. PMID 33355350
- [Background] Rubin LG, Levin MJ, Ljungman P, Davies EG, Avery R, Tomblyn M, Bousvaros A, Dhanireddy S, Sung L, Keyserling H, Kang I; Infectious Diseases Society of America. 2013 IDSA clinical practice guideline for vaccination of the immunocompromised host. Clin Infect Dis. 2014 Feb;58(3):309-18. doi: 10.1093/cid/cit816. PMID 24421306
- [Background] Im Y, Kang D, Ko RE, Lee YJ, Lim SY, Park S, Na SJ, Chung CR, Park MH, Oh DK, Lim CM, Suh GY; Korean Sepsis Alliance (KSA) investigators. Time-to-antibiotics and clinical outcomes in patients with sepsis and septic shock: a prospective nationwide multicenter cohort study. Crit Care. 2022 Jan 13;26(1):19. doi: 10.1186/s13054-021-03883-0. PMID 35027073
- [Background] Taylor SP, Kowalkowski MA, Skewes S, Chou SH. Real-World Implications of Updated Surviving Sepsis Campaign Antibiotic Timing Recommendations. Crit Care Med. 2024 Jul 1;52(7):1002-1006. doi: 10.1097/CCM.0000000000006240. Epub 2024 Feb 22. PMID 38385751
- [Background] Rose N, Matthaus-Kramer C, Schwarzkopf D, Scherag A, Born S, Reinhart K, Fleischmann-Struzek C. Association between sepsis incidence and regional socioeconomic deprivation and health care capacity in Germany - an ecological study. BMC Public Health. 2021 Sep 7;21(1):1636. doi: 10.1186/s12889-021-11629-4. PMID 34493250
- [Background] Cornistein W, Santonato D, Novau PA, Fabbro LG, Jorge MF, Malvicini MA, Vilches V, Iudica FM. Synergy between infection control and antimicrobial stewardship programs to control carbapenem-resistant Enterobacterales. Antimicrob Steward Healthc Epidemiol. 2023 Sep 26;3(1):e162. doi: 10.1017/ash.2023.439. eCollection 2023. PMID 37771737
- [Background] Kherabi Y, Thy M, Bouzid D, Antcliffe DB, Rawson TM, Peiffer-Smadja N. Machine learning to predict antimicrobial resistance: future applications in clinical practice? Infect Dis Now. 2024 Apr;54(3):104864. doi: 10.1016/j.idnow.2024.104864. Epub 2024 Feb 12. PMID 38355048
- [Background] Peiffer-Smadja N, Delliere S, Rodriguez C, Birgand G, Lescure FX, Fourati S, Ruppe E. Machine learning in the clinical microbiology laboratory: has the time come for routine practice? Clin Microbiol Infect. 2020 Oct;26(10):1300-1309. doi: 10.1016/j.cmi.2020.02.006. Epub 2020 Feb 12. PMID 32061795
- [Background] Bisarya R, Song X, Salle J, Liu M, Patel A, Simpson SQ. Antibiotic Timing and Progression to Septic Shock Among Patients in the ED With Suspected Infection. Chest. 2022 Jan;161(1):112-120. doi: 10.1016/j.chest.2021.06.029. Epub 2021 Jun 26. PMID 34186038
- [Background] Mertz D, Frei R, Periat N, Zimmerli M, Battegay M, Fluckiger U, Widmer AF. Exclusive Staphylococcus aureus throat carriage: at-risk populations. Arch Intern Med. 2009 Jan 26;169(2):172-8. doi: 10.1001/archinternmed.2008.536. PMID 19171814
- [Background] Giannella M, Trecarichi EM, De Rosa FG, Del Bono V, Bassetti M, Lewis RE, Losito AR, Corcione S, Saffioti C, Bartoletti M, Maiuro G, Cardellino CS, Tedeschi S, Cauda R, Viscoli C, Viale P, Tumbarello M. Risk factors for carbapenem-resistant Klebsiella pneumoniae bloodstream infection among rectal carriers: a prospective observational multicentre study. Clin Microbiol Infect. 2014 Dec;20(12):1357-62. doi: 10.1111/1469-0691.12747. Epub 2014 Aug 11. PMID 24980276
- [Background] Cano A, Gutierrez-Gutierrez B, Machuca I, Torre-Gimenez J, Gracia-Ahufinger I, Natera AM, Perez-Nadales E, Caston JJ, Rodriguez-Bano J, Martinez-Martinez L, Torre-Cisneros J. Association between Timing of Colonization and Risk of Developing Klebsiella pneumoniae Carbapenemase-Producing K. pneumoniae Infection in Hospitalized Patients. Microbiol Spectr. 2022 Apr 27;10(2):e0197021. doi: 10.1128/spectrum.01970-21. Epub 2022 Mar 24. PMID 35323035
- [Background] Temkin E, Solter E, Lugassy C, Chen D, Cohen A, Schwaber MJ, Carmeli Y; CPE Working Group. The Natural History of Carbapenemase-Producing Enterobacterales: Progression From Carriage of Various Carbapenemases to Bloodstream Infection. Clin Infect Dis. 2024 Jul 19;79(1):22-29. doi: 10.1093/cid/ciae110. PMID 38447961
- [Background] Blagojevic C, Brown KA, Diong C, Fridman DJ, Johnstone J, Langford BJ, Lee SM, MacFadden DR, Schwartz KL, Daneman N. Long-term Risk of Infection Among Patients Colonized With Antimicrobial-Resistant Pathogens: A Population-wide Cohort Study. Open Forum Infect Dis. 2024 Dec 2;11(12):ofae712. doi: 10.1093/ofid/ofae712. eCollection 2024 Dec. PMID 39703788
- [Background] Schlebusch S, Graham RMA, Jennison AV, Lassig-Smith MM, Harris PNA, Lipman J, O Cuiv P, Paterson DL. Standard rectal swabs as a surrogate sample for gut microbiome monitoring in intensive care. BMC Microbiol. 2022 Apr 12;22(1):99. doi: 10.1186/s12866-022-02487-0. PMID 35413802
- [Background] Tumbarello M, Trecarichi EM, Bassetti M, De Rosa FG, Spanu T, Di Meco E, Losito AR, Parisini A, Pagani N, Cauda R. Identifying patients harboring extended-spectrum-beta-lactamase-producing Enterobacteriaceae on hospital admission: derivation and validation of a scoring system. Antimicrob Agents Chemother. 2011 Jul;55(7):3485-90. doi: 10.1128/AAC.00009-11. Epub 2011 May 2. PMID 21537020
- [Background] Blot S, Antonelli M, Arvaniti K, Blot K, Creagh-Brown B, de Lange D, De Waele J, Deschepper M, Dikmen Y, Dimopoulos G, Eckmann C, Francois G, Girardis M, Koulenti D, Labeau S, Lipman J, Lipovestky F, Maseda E, Montravers P, Mikstacki A, Paiva JA, Pereyra C, Rello J, Timsit JF, Vogelaers D; Abdominal Sepsis Study (AbSeS) group on behalf of the Trials Group of the European Society of Intensive Care Medicine. Epidemiology of intra-abdominal infection and sepsis in critically ill patients: "AbSeS", a multinational observational cohort study and ESICM Trials Group Project. Intensive Care Med. 2019 Dec;45(12):1703-1717. doi: 10.1007/s00134-019-05819-3. Epub 2019 Oct 29. PMID 31664501
- [Background] Bassetti M, Righi E, Vena A, Graziano E, Russo A, Peghin M. Risk stratification and treatment of ICU-acquired pneumonia caused by multidrug- resistant/extensively drug-resistant/pandrug-resistant bacteria. Curr Opin Crit Care. 2018 Oct;24(5):385-393. doi: 10.1097/MCC.0000000000000534. PMID 30156569
- [Background] De Waele JJ, Boelens J, Leroux-Roels I. Multidrug-resistant bacteria in ICU: fact or myth. Curr Opin Anaesthesiol. 2020 Apr;33(2):156-161. doi: 10.1097/ACO.0000000000000830. PMID 31904697
- [Background] Pea F, Viale P. The antimicrobial therapy puzzle: could pharmacokinetic-pharmacodynamic relationships be helpful in addressing the issue of appropriate pneumonia treatment in critically ill patients? Clin Infect Dis. 2006 Jun 15;42(12):1764-71. doi: 10.1086/504383. Epub 2006 May 10. PMID 16705585
- [Background] Echegorry M, Marchetti P, Sanchez C, Olivieri L, Faccone D, Martino F, Sarkis Badola T, Ceriana P, Rapoport M, Lucero C, Albornoz E, Recapt-Ar Group, Corso A, Pasteran F. National Multicenter Study on the Prevalence of Carbapenemase-Producing Enterobacteriaceae in the Post-COVID-19 Era in Argentina: The RECAPT-AR Study. Antibiotics (Basel). 2024 Nov 27;13(12):1139. doi: 10.3390/antibiotics13121139. PMID 39766529
- [Background] Lee YL, Ko WC, Hsueh PR. Geographic patterns of global isolates of carbapenem-resistant Klebsiella pneumoniae and the activity of ceftazidime/avibactam, meropenem/vaborbactam, and comparators against these isolates: Results from the Antimicrobial Testing Leadership and Surveillance (ATLAS) program, 2020. Int J Antimicrob Agents. 2022 Nov-Dec;60(5-6):106679. doi: 10.1016/j.ijantimicag.2022.106679. Epub 2022 Oct 12. PMID 36241011
- [Background] Thomas GR, Corso A, Pasteran F, Shal J, Sosa A, Pillonetto M, de Souza Peral RT, Hormazabal JC, Araya P, Saavedra SY, Ovalle MV, Jimenez Pearson MA, Chacon GC, Carbon E, Mazariegos Herrera CJ, Velasquez SDCG, Satan-Salazar C, Villavicencio F, Touchet NM, Busignani S, Mayta-Barrios M, Ramirez-Illescas J, Vega ML, Mogdasy C, Rosas V, Salgado N, Quiroz R, El-Omeiri N, Galas MF, Ramon-Pardo P, Melano RG. Increased Detection of Carbapenemase-Producing Enterobacterales Bacteria in Latin America and the Caribbean during the COVID-19 Pandemic. Emerg Infect Dis. 2022 Nov;28(11):1-8. doi: 10.3201/eid2811.220415. PMID 36286547
- [Background] Potter RF, D'Souza AW, Dantas G. The rapid spread of carbapenem-resistant Enterobacteriaceae. Drug Resist Updat. 2016 Nov;29:30-46. doi: 10.1016/j.drup.2016.09.002. Epub 2016 Sep 19. PMID 27912842
- [Background] Livermore DM, Nicolau DP, Hopkins KL, Meunier D. Carbapenem-Resistant Enterobacterales, Carbapenem Resistant Organisms, Carbapenemase-Producing Enterobacterales, and Carbapenemase-Producing Organisms: Terminology Past its "Sell-By Date" in an Era of New Antibiotics and Regional Carbapenemase Epidemiology. Clin Infect Dis. 2020 Oct 23;71(7):1776-1782. doi: 10.1093/cid/ciaa122. PMID 32025698
- [Background] Tamma PD, Doi Y, Bonomo RA, Johnson JK, Simner PJ; Antibacterial Resistance Leadership Group. A Primer on AmpC beta-Lactamases: Necessary Knowledge for an Increasingly Multidrug-resistant World. Clin Infect Dis. 2019 Sep 27;69(8):1446-1455. doi: 10.1093/cid/ciz173. PMID 30838380
- [Background] Osano E, Arakawa Y, Wacharotayankun R, Ohta M, Horii T, Ito H, Yoshimura F, Kato N. Molecular characterization of an enterobacterial metallo beta-lactamase found in a clinical isolate of Serratia marcescens that shows imipenem resistance. Antimicrob Agents Chemother. 1994 Jan;38(1):71-8. doi: 10.1128/AAC.38.1.71. PMID 8141584
- [Background] Lauretti L, Riccio ML, Mazzariol A, Cornaglia G, Amicosante G, Fontana R, Rossolini GM. Cloning and characterization of blaVIM, a new integron-borne metallo-beta-lactamase gene from a Pseudomonas aeruginosa clinical isolate. Antimicrob Agents Chemother. 1999 Jul;43(7):1584-90. doi: 10.1128/AAC.43.7.1584. PMID 10390207
- [Background] Yong D, Toleman MA, Giske CG, Cho HS, Sundman K, Lee K, Walsh TR. Characterization of a new metallo-beta-lactamase gene, bla(NDM-1), and a novel erythromycin esterase gene carried on a unique genetic structure in Klebsiella pneumoniae sequence type 14 from India. Antimicrob Agents Chemother. 2009 Dec;53(12):5046-54. doi: 10.1128/AAC.00774-09. Epub 2009 Sep 21. PMID 19770275
- [Background] Martinez-Martinez L, Gonzalez-Lopez JJ. Carbapenemases in Enterobacteriaceae: types and molecular epidemiology. Enferm Infecc Microbiol Clin. 2014 Dec;32 Suppl 4:4-9. doi: 10.1016/S0213-005X(14)70168-5. PMID 25542046
- [Background] Sawa T, Kooguchi K, Moriyama K. Molecular diversity of extended-spectrum beta-lactamases and carbapenemases, and antimicrobial resistance. J Intensive Care. 2020 Jan 28;8:13. doi: 10.1186/s40560-020-0429-6. eCollection 2020. PMID 32015881
- [Background] Sati H, Carrara E, Savoldi A, Hansen P, Garlasco J, Campagnaro E, Boccia S, Castillo-Polo JA, Magrini E, Garcia-Vello P, Wool E, Gigante V, Duffy E, Cassini A, Huttner B, Pardo PR, Naghavi M, Mirzayev F, Zignol M, Cameron A, Tacconelli E; WHO Bacterial Priority Pathogens List Advisory Group. The WHO Bacterial Priority Pathogens List 2024: a prioritisation study to guide research, development, and public health strategies against antimicrobial resistance. Lancet Infect Dis. 2025 Sep;25(9):1033-1043. doi: 10.1016/S1473-3099(25)00118-5. Epub 2025 Apr 14. PMID 40245910
- [Background] Zhou R, Fang X, Zhang J, Zheng X, Shangguan S, Chen S, Shen Y, Liu Z, Li J, Zhang R, Shen J, Walsh TR, Wang Y. Impact of carbapenem resistance on mortality in patients infected with Enterobacteriaceae: a systematic review and meta-analysis. BMJ Open. 2021 Dec 14;11(12):e054971. doi: 10.1136/bmjopen-2021-054971. PMID 34907071
- [Background] van Duin D, Doi Y. The global epidemiology of carbapenemase-producing Enterobacteriaceae. Virulence. 2017 May 19;8(4):460-469. doi: 10.1080/21505594.2016.1222343. Epub 2016 Aug 11. PMID 27593176
- [Background] Winiszewski H, Despres C, Puyraveau M, Lagoutte-Renosi J, Montange D, Besch G, Floury SP, Chaignat C, Labro G, Vettoretti L, Clairet AL, Capellier G, Vivet B, Piton G. beta-lactam dosing at the early phase of sepsis: Performance of a pragmatic protocol for target concentration achievement in a prospective cohort study. J Crit Care. 2022 Feb;67:141-146. doi: 10.1016/j.jcrc.2021.10.023. Epub 2021 Nov 9. PMID 34768176
- [Background] Li X, Jiang Z. Do prolonged infusions of beta-lactam antibiotics improve outcomes in critically ill patients with sepsis? It is time to say yes. Crit Care. 2024 Nov 21;28(1):380. doi: 10.1186/s13054-024-05139-z. No abstract available. PMID 39574173
- [Background] Shappell CN, Klompas M, Rhee C. Do Prolonged Infusions of beta-Lactam Antibiotics Improve Outcomes in Critically Ill Patients With Sepsis? JAMA. 2023 Jul 11;330(2):126-128. doi: 10.1001/jama.2023.6483. No abstract available. PMID 37326478
- [Background] Cusack R, Little E, Martin-Loeches I. Practical Lessons on Antimicrobial Therapy for Critically Ill Patients. Antibiotics (Basel). 2024 Feb 6;13(2):162. doi: 10.3390/antibiotics13020162. PMID 38391547
- [Background] Roberts JA, Taccone FS, Lipman J. Understanding PK/PD. Intensive Care Med. 2016 Nov;42(11):1797-1800. doi: 10.1007/s00134-015-4032-6. Epub 2015 Sep 3. No abstract available. PMID 26334756
- [Background] Khilnani GC, Zirpe K, Hadda V, Mehta Y, Madan K, Kulkarni A, Mohan A, Dixit S, Guleria R, Bhattacharya P. Guidelines for Antibiotic Prescription in Intensive Care Unit. Indian J Crit Care Med. 2019 Jan;23(Suppl 1):S1-S63. doi: 10.5005/jp-journals-10071-23101. PMID 31516211
- [Background] Rhee C, Kadri SS, Dekker JP, Danner RL, Chen HC, Fram D, Zhang F, Wang R, Klompas M; CDC Prevention Epicenters Program. Prevalence of Antibiotic-Resistant Pathogens in Culture-Proven Sepsis and Outcomes Associated With Inadequate and Broad-Spectrum Empiric Antibiotic Use. JAMA Netw Open. 2020 Apr 1;3(4):e202899. doi: 10.1001/jamanetworkopen.2020.2899. PMID 32297949
- [Background] Larsson DGJ, Flach CF. Antibiotic resistance in the environment. Nat Rev Microbiol. 2022 May;20(5):257-269. doi: 10.1038/s41579-021-00649-x. Epub 2021 Nov 4. PMID 34737424
- [Background] Santacroce L, Di Domenico M, Montagnani M, Jirillo E. Antibiotic Resistance and Microbiota Response. Curr Pharm Des. 2023;29(5):356-364. doi: 10.2174/1381612829666221219093450. PMID 36537602
- [Background] De Bus L, Depuydt P, Steen J, Dhaese S, De Smet K, Tabah A, Akova M, Cotta MO, De Pascale G, Dimopoulos G, Fujitani S, Garnacho-Montero J, Leone M, Lipman J, Ostermann M, Paiva JA, Schouten J, Sjovall F, Timsit JF, Roberts JA, Zahar JR, Zand F, Zirpe K, De Waele JJ; DIANA study group. Antimicrobial de-escalation in the critically ill patient and assessment of clinical cure: the DIANA study. Intensive Care Med. 2020 Jul;46(7):1404-1417. doi: 10.1007/s00134-020-06111-5. Epub 2020 Jun 9. PMID 32519003
- [Background] Teshome BF, Park T, Arackal J, Hampton N, Kollef MH, Micek ST. Preventing New Gram-negative Resistance Through Beta-lactam De-escalation in Hospitalized Patients With Sepsis: A Retrospective Cohort Study. Clin Infect Dis. 2024 Oct 15;79(4):826-833. doi: 10.1093/cid/ciae253. PMID 38842541
- [Background] Spellberg B, Rice LB. Duration of Antibiotic Therapy: Shorter Is Better. Ann Intern Med. 2019 Aug 6;171(3):210-211. doi: 10.7326/M19-1509. Epub 2019 Jul 9. No abstract available. PMID 31284302
- [Background] Rhee C, Filbin M, Klompas M. Measuring Diagnostic Accuracy for Infection in Patients Treated for Sepsis: An Important but Challenging Exercise. Clin Infect Dis. 2023 Jun 16;76(12):2056-2058. doi: 10.1093/cid/ciad105. No abstract available. PMID 36804679
- [Background] Arulkumaran N, Routledge M, Schlebusch S, Lipman J, Conway Morris A. Antimicrobial-associated harm in critical care: a narrative review. Intensive Care Med. 2020 Feb;46(2):225-235. doi: 10.1007/s00134-020-05929-3. Epub 2020 Jan 29. PMID 31996961
- [Background] Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CG, Harbarth S, Hindler JF, Kahlmeter G, Olsson-Liljequist B, Paterson DL, Rice LB, Stelling J, Struelens MJ, Vatopoulos A, Weber JT, Monnet DL. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect. 2012 Mar;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x. Epub 2011 Jul 27. PMID 21793988
- [Background] GBD 2021 Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance 1990-2021: a systematic analysis with forecasts to 2050. Lancet. 2024 Sep 28;404(10459):1199-1226. doi: 10.1016/S0140-6736(24)01867-1. Epub 2024 Sep 16. PMID 39299261
- [Background] Coluzzi C, Rocha EPC. The Spread of Antibiotic Resistance Is Driven by Plasmids Among the Fastest Evolving and of Broadest Host Range. Mol Biol Evol. 2025 Mar 5;42(3):msaf060. doi: 10.1093/molbev/msaf060. PMID 40098486
- [Background] Bharadwaj A, Rastogi A, Pandey S, Gupta S, Sohal JS. Multidrug-Resistant Bacteria: Their Mechanism of Action and Prophylaxis. Biomed Res Int. 2022 Sep 5;2022:5419874. doi: 10.1155/2022/5419874. eCollection 2022. PMID 36105930
- [Background] Aslam B, Khurshid M, Arshad MI, Muzammil S, Rasool M, Yasmeen N, Shah T, Chaudhry TH, Rasool MH, Shahid A, Xueshan X, Baloch Z. Antibiotic Resistance: One Health One World Outlook. Front Cell Infect Microbiol. 2021 Nov 25;11:771510. doi: 10.3389/fcimb.2021.771510. eCollection 2021. PMID 34900756
- [Background] Conde KA, Silva E, Silva CO, Ferreira E, Freitas FG, Castro I, Rea-Neto A, Grion CM, Moura AD, Lobo SM, Azevedo LC, Machado FR. Differences in sepsis treatment and outcomes between public and private hospitals in Brazil: a multicenter observational study. PLoS One. 2013 Jun 6;8(6):e64790. doi: 10.1371/journal.pone.0064790. Print 2013. PMID 23762255
- [Background] Arefian H, Heublein S, Scherag A, Brunkhorst FM, Younis MZ, Moerer O, Fischer D, Hartmann M. Hospital-related cost of sepsis: A systematic review. J Infect. 2017 Feb;74(2):107-117. doi: 10.1016/j.jinf.2016.11.006. Epub 2016 Nov 21. PMID 27884733
- [Background] Buchman TG, Simpson SQ, Sciarretta KL, Finne KP, Sowers N, Collier M, Chavan S, Oke I, Pennini ME, Santhosh A, Wax M, Woodbury R, Chu S, Merkeley TG, Disbrow GL, Bright RA, MaCurdy TE, Kelman JA. Sepsis Among Medicare Beneficiaries: 1. The Burdens of Sepsis, 2012-2018. Crit Care Med. 2020 Mar;48(3):276-288. doi: 10.1097/CCM.0000000000004224. PMID 32058366
- [Background] Paoli CJ, Reynolds MA, Sinha M, Gitlin M, Crouser E. Epidemiology and Costs of Sepsis in the United States-An Analysis Based on Timing of Diagnosis and Severity Level. Crit Care Med. 2018 Dec;46(12):1889-1897. doi: 10.1097/CCM.0000000000003342. PMID 30048332
- [Background] Wang T, Derhovanessian A, De Cruz S, Belperio JA, Deng JC, Hoo GS. Subsequent infections in survivors of sepsis: epidemiology and outcomes. J Intensive Care Med. 2014 Mar-Apr;29(2):87-95. doi: 10.1177/0885066612467162. Epub 2012 Dec 26. PMID 23753224
- [Background] van der Slikke EC, An AY, Hancock REW, Bouma HR. Exploring the pathophysiology of post-sepsis syndrome to identify therapeutic opportunities. EBioMedicine. 2020 Nov;61:103044. doi: 10.1016/j.ebiom.2020.103044. Epub 2020 Oct 8. PMID 33039713
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Schultz MJ, Dunser MW, Dondorp AM, Adhikari NK, Iyer S, Kwizera A, Lubell Y, Papali A, Pisani L, Riviello BD, Angus DC, Azevedo LC, Baker T, Diaz JV, Festic E, Haniffa R, Jawa R, Jacob ST, Kissoon N, Lodha R, Martin-Loeches I, Lundeg G, Misango D, Mer M, Mohanty S, Murthy S, Musa N, Nakibuuka J, Serpa Neto A, Nguyen Thi Hoang M, Nguyen Thien B, Pattnaik R, Phua J, Preller J, Povoa P, Ranjit S, Talmor D, Thevanayagam J, Thwaites CL; Global Intensive Care Working Group of the European Society of Intensive Care Medicine. Current challenges in the management of sepsis in ICUs in resource-poor settings and suggestions for the future. Intensive Care Med. 2017 May;43(5):612-624. doi: 10.1007/s00134-017-4750-z. Epub 2017 Mar 27. PMID 28349179
- [Background] Thwaites CL, Lundeg G, Dondorp AM; sepsis in resource-limited settings-expert consensus recommendations group of the European Society of Intensive Care Medicine (ESICM) and the Mahidol-Oxford Research Unit (MORU) in Bangkok, Thailand. Recommendations for infection management in patients with sepsis and septic shock in resource-limited settings. Intensive Care Med. 2016 Dec;42(12):2040-2042. doi: 10.1007/s00134-016-4415-3. Epub 2016 Jun 21. No abstract available. PMID 27324344
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Levy MM, Rhodes A, Phillips GS, Townsend SR, Schorr CA, Beale R, Osborn T, Lemeshow S, Chiche JD, Artigas A, Dellinger RP. Surviving Sepsis Campaign: association between performance metrics and outcomes in a 7.5-year study. Crit Care Med. 2015 Jan;43(1):3-12. doi: 10.1097/CCM.0000000000000723. PMID 25275252
- [Background] Machado FR, Cavalcanti AB, Bozza FA, Ferreira EM, Angotti Carrara FS, Sousa JL, Caixeta N, Salomao R, Angus DC, Pontes Azevedo LC; SPREAD Investigators; Latin American Sepsis Institute Network. The epidemiology of sepsis in Brazilian intensive care units (the Sepsis PREvalence Assessment Database, SPREAD): an observational study. Lancet Infect Dis. 2017 Nov;17(11):1180-1189. doi: 10.1016/S1473-3099(17)30322-5. Epub 2017 Aug 17. PMID 28826588
- [Background] Divatia JV, Amin PR, Ramakrishnan N, Kapadia FN, Todi S, Sahu S, Govil D, Chawla R, Kulkarni AP, Samavedam S, Jani CK, Rungta N, Samaddar DP, Mehta S, Venkataraman R, Hegde A, Bande BD, Dhanuka S, Singh V, Tewari R, Zirpe K, Sathe P; INDICAPS Study Investigators. Intensive Care in India: The Indian Intensive Care Case Mix and Practice Patterns Study. Indian J Crit Care Med. 2016 Apr;20(4):216-25. doi: 10.4103/0972-5229.180042. PMID 27186054
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Shankar-Hari M, Harrison DA, Rowan KM. Differences in Impact of Definitional Elements on Mortality Precludes International Comparisons of Sepsis Epidemiology-A Cohort Study Illustrating the Need for Standardized Reporting. Crit Care Med. 2016 Dec;44(12):2223-2230. doi: 10.1097/CCM.0000000000001876. PMID 27352126
- [Background] Liu V, Escobar GJ, Greene JD, Soule J, Whippy A, Angus DC, Iwashyna TJ. Hospital deaths in patients with sepsis from 2 independent cohorts. JAMA. 2014 Jul 2;312(1):90-2. doi: 10.1001/jama.2014.5804. No abstract available. PMID 24838355
- [Background] Weng L, Xu Y, Yin P, Wang Y, Chen Y, Liu W, Li S, Peng JM, Dong R, Hu XY, Jiang W, Wang CY, Gao P, Zhou MG, Du B; China Critical Care Clinical Trials Group (CCCCTG). National incidence and mortality of hospitalized sepsis in China. Crit Care. 2023 Mar 4;27(1):84. doi: 10.1186/s13054-023-04385-x. PMID 36870989
- [Background] Southeast Asia Infectious Disease Clinical Research Network. Causes and outcomes of sepsis in southeast Asia: a multinational multicentre cross-sectional study. Lancet Glob Health. 2017 Feb;5(2):e157-e167. doi: 10.1016/S2214-109X(17)30007-4. PMID 28104185
- [Background] Fleischmann-Struzek C, Mikolajetz A, Schwarzkopf D, Cohen J, Hartog CS, Pletz M, Gastmeier P, Reinhart K. Challenges in assessing the burden of sepsis and understanding the inequalities of sepsis outcomes between National Health Systems: secular trends in sepsis and infection incidence and mortality in Germany. Intensive Care Med. 2018 Nov;44(11):1826-1835. doi: 10.1007/s00134-018-5377-4. Epub 2018 Oct 4. PMID 30284637
- [Background] Rhee C, Dantes R, Epstein L, Murphy DJ, Seymour CW, Iwashyna TJ, Kadri SS, Angus DC, Danner RL, Fiore AE, Jernigan JA, Martin GS, Septimus E, Warren DK, Karcz A, Chan C, Menchaca JT, Wang R, Gruber S, Klompas M; CDC Prevention Epicenter Program. Incidence and Trends of Sepsis in US Hospitals Using Clinical vs Claims Data, 2009-2014. JAMA. 2017 Oct 3;318(13):1241-1249. doi: 10.1001/jama.2017.13836. PMID 28903154
- [Background] La Via L, Sangiorgio G, Stefani S, Marino A, Nunnari G, Cocuzza S, La Mantia I, Cacopardo B, Stracquadanio S, Spampinato S, Lavalle S, Maniaci A. The Global Burden of Sepsis and Septic Shock. Epidemiologia (Basel). 2024 Jul 25;5(3):456-478. doi: 10.3390/epidemiologia5030032. PMID 39189251
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Kumar NR, Balraj TA, Kempegowda SN, Prashant A. Multidrug-Resistant Sepsis: A Critical Healthcare Challenge. Antibiotics (Basel). 2024 Jan 4;13(1):46. doi: 10.3390/antibiotics13010046. PMID 38247605
- [Background] Velazquez-Meza ME, Galarde-Lopez M, Carrillo-Quiroz B, Alpuche-Aranda CM. Antimicrobial resistance: One Health approach. Vet World. 2022 Mar;15(3):743-749. doi: 10.14202/vetworld.2022.743-749. Epub 2022 Mar 28. PMID 35497962
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Ramasco F, Mendez R, Suarez de la Rica A, Gonzalez de Castro R, Maseda E. Sepsis Stewardship: The Puzzle of Antibiotic Therapy in the Context of Individualization of Decision Making. J Pers Med. 2024 Jan 18;14(1):106. doi: 10.3390/jpm14010106. PMID 38248807
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Muteeb G, Rehman MT, Shahwan M, Aatif M. Origin of Antibiotics and Antibiotic Resistance, and Their Impacts on Drug Development: A Narrative Review. Pharmaceuticals (Basel). 2023 Nov 15;16(11):1615. doi: 10.3390/ph16111615. PMID 38004480
- [Background] Llor C, Bjerrum L. Antimicrobial resistance: risk associated with antibiotic overuse and initiatives to reduce the problem. Ther Adv Drug Saf. 2014 Dec;5(6):229-41. doi: 10.1177/2042098614554919. PMID 25436105
- See also: CDC. About. In: Sepsis [Internet]. 13 May 2024 [cited 9 Mar 2025]. Available: https://www.cdc.gov/sepsis/about/index.html — https://www.cdc.gov/sepsis/about/index.html
- See also: One Health. [cited 22 Mar 2025]. Available: https://www.who.int/europe/initiatives/one-health — https://www.who.int/europe/initiatives/one-health
- See also: References & Sources. In: The UK Sepsis Trust [Internet]. 9 Aug 2024 [cited 9 Mar 2025]. Available: https://sepsistrust.org/about-sepsis/references-sources/ — https://sepsistrust.org/about-sepsis/references-sources/
- See also: Surviving Sepsis Campaign. In: Society of Critical Care Medicine (SCCM) [Internet]. [cited 6 Apr 2025]. Available: https://www.sccm.org/survivingsepsiscampaign — https://www.sccm.org/survivingsepsiscampaign
- See also: Global antimicrobial resistance and use surveillance system (GLASS) report: 2022. World Health Organization; 9 Dec 2022 [cited 3 Oct 2023]. Available: https://www.who.int/publications/i/item/9789240062702 — https://www.who.int/publications/i/item/9789240062702
- See also: Bastin MT, Rech M, Betthauser K, Heavner M, Horng M, King T, et al. 1206: Beta-lactam dosing in patients with sepsis and Aki: A multicenter observational study. Crit Care Med. 2023;51: 601-601. — https://journals.lww.com/ccmjournal/citation/2023/01001/1206__beta_lactam_dosing_in_patients_with_sepsis.1173.aspx
- See also: Surveillance of antimicrobial resistance in Europe 2017. In: European Centre for Disease Prevention and Control [Internet]. 15 Nov 2018 [cited 3 Oct 2023]. Available: https://www.ecdc.europa.eu/en/publications-data/surveillance-antimicrobial-resistance-e — https://www.ecdc.europa.eu/en/publications-data/surveillance-antimicrobial-resistance-europe-2017
- See also: INFECCIONES DE PIEL Y PARTES BLANDAS Y PREVALENCIA DE SAMR EN PACIENTES AMBULATORIOS EN UN HOSPITAL GENERAL DE CABA. [cited 8 Mar 2025]. Available: https://infectologia.info/abstracts/infecciones-de-piel-y-partes-blandas-y-prevalencia-de-samr-en-paciente — https://infectologia.info/abstracts/infecciones-de-piel-y-partes-blandas-y-prevalencia-de-samr-en-pacientes-ambulatorios-en-un-hospital-general-de-caba/
- See also: [No title]. [cited 8 Mar 2025]. Available: http://antimicrobianos.com.ar/wp-content/uploads/2023/10/Mapas-de-Resistencia-Antimicrobiana-Red-WHONET-Argentina-2022.pdf — http://antimicrobianos.com.ar/wp-content/uploads/2023/10/Mapas-de-Resistencia-Antimicrobiana-Red-WHONET-Argentina-2022.pdf
- See also: Nov. INFORME RESISTENCIA 2023 - ARGENTINA. [cited 24 Mar 2025]. Available: http://antimicrobianos.com.ar/2024/11/informe-resistencia-2023-argentina/ — http://antimicrobianos.com.ar/2024/11/informe-resistencia-2023-argentina/
- See also: Fosch S, Yones C, Trossero M, Grosso O, Nepote A. Portación nasal de Staphylococcus aureus en individuos de la comunidad: factores epidemiológicos. Acta bioquím clín latinoam. 2012;46: 59-68. — https://www.scielo.org.ar/scielo.php?script=sci_arttext&pid=S0325-29572012000100009
- See also: THE 17 GOALS. [cited 13 Apr 2025]. Available: https://sdgs.un.org/goals — https://sdgs.un.org/goals
- See also: Goal 3. [cited 13 Apr 2025]. Available: https://sdgs.un.org/goals/goal3 — https://sdgs.un.org/goals/goal3
- See also: Objetivo 9. [cited 14 Apr 2025]. Available: https://sdgs.un.org/es/goals/goal9 — https://sdgs.un.org/es/goals/goal9
- See also: Goal 10. [cited 13 Apr 2025]. Available: https://sdgs.un.org/goals/goal10 — https://sdgs.un.org/goals/goal10
- See also: Ratti MFG, Martinez B. Reestructuración de la Central de Emergencias durante la pandemia. Rev Hosp Ital BAires. 2022;42: 46-48. — https://ojs.hospitalitaliano.org.ar/index.php/revistahi/article/view/147
- See also: [No title]. [cited 16 Apr 2025]. Available: https://hiba.hospitalitaliano.org.ar/archivos/noticias_archivos/74/archivos/Plan%20de%20Accion%20Central%20de%20Emergencias%20-%20Covid19.pdf — https://hiba.hospitalitaliano.org.ar/archivos/noticias_archivos/74/archivos/Plan%20de%20Accion%20Central%20de%20Emergencias%20-%20Covid19.pdf
- See also: [No title]. [cited 16 Apr 2025]. Available: https://faso.org.ar/imagenes/covid/protocolo_italiano-17-4.pdf — https://faso.org.ar/imagenes/covid/protocolo_italiano-17-4.pdf
- See also: Centro Nacional de Terminología en Salud. In: Argentina.gob.ar [Internet]. 19 Jul 2021 [cited 12 Nov 2023]. Available: https://www.argentina.gob.ar/salud/terminologia — https://www.argentina.gob.ar/salud/terminologia
- See also: [No title]. [cited 16 Apr 2025]. Available: https://www.hospitalitaliano.org.ar/multimedia/archivos/noticias_archivos/109/guias_para_medicos/109_sepsis.pdf — https://www.hospitalitaliano.org.ar/multimedia/archivos/noticias_archivos/109/guias_para_medicos/109_sepsis.pdf
- See also: [No title]. [cited 16 Apr 2025]. Available: https://hiba.hospitalitaliano.org.ar/archivos/noticias_archivos/109/archivos/Sepsis%20sitio%20infecto%20final-converted.pdf — https://hiba.hospitalitaliano.org.ar/archivos/noticias_archivos/109/archivos/Sepsis%20sitio%20infecto%20final-converted.pdf
- See also: El Gobierno Nacional decretó el aislamiento social preventivo y obligatorio. In: Argentina.gob.ar [Internet]. 20 Mar 2020 [cited 14 Apr 2025]. Available: https://www.argentina.gob.ar/noticias/el-gobierno-nacional-decreto-el-aislamiento-social-preventivo- — https://www.argentina.gob.ar/noticias/el-gobierno-nacional-decreto-el-aislamiento-social-preventivo-y-obligatorio
- See also: Sep. AÑO 2023. [cited 13 Apr 2025]. Available: http://antimicrobianos.com.ar/2024/09/2023/ — http://antimicrobianos.com.ar/2024/09/2023/
- See also: [No title]. [cited 13 Apr 2025]. Available: http://antimicrobianos.com.ar/wp-content/uploads/2024/12/Mapas-de-Resistencia-Antimicrobiana-Red-WHONET-Argentina-2023.pdf — http://antimicrobianos.com.ar/wp-content/uploads/2024/12/Mapas-de-Resistencia-Antimicrobiana-Red-WHONET-Argentina-2023.pdf
- See also: Immunocompromised Travelers. [cited 18 Feb 2025]. Available: https://wwwnc.cdc.gov/travel/yellowbook/2024/additional-considerations/immunocompromised-travelers — https://wwwnc.cdc.gov/travel/yellowbook/2024/additional-considerations/immunocompromised-travelers
- See also: [No title]. [cited 11 Feb 2024]. Available: https://www.sah.org.ar/revistasah/numeros/vol21/extra3/36-vol21-extra_noviembre.pdf — https://www.sah.org.ar/revistasah/numeros/vol21/extra3/36-vol21-extra_noviembre.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT07167173/Prot_SAP_000.pdf